CLINICAL TRIAL: NCT07260890
Title: Diagnostic Accuracy of Stroke Volume Variation (SVV) vs Pleth Variability Index (PVI) for Predicting Fluid Responsiveness in Laparoscopic Major Abdominal Surgery-A Prospective, Paired, Cohort Study
Brief Title: Paired Comparison of SVV and PVI Accuracy
Status: Recruiting | Type: Observational
Sponsor: Wonkwang University Hospital (Other)
Responsible Party: Principal Investigator, Cheol Lee,MD,PhD,, Professor, Wonkwang University Hospital
Other Study IDs: Wonkwang UH 22
Record Dates: First submitted 2025-11-13; First posted 2025-12-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Perioperative Care; Fluid Therapy; Monitoring, Physiologic; Hemodynamics; Laparoscopy
Keywords: stroke volume variation; SVV; Pleth Variability Index; PVI; fluid responsiveness; goal-directed fluid therapy; GDFT; pneumoperitoneum; diagnostic accuracy; ROC; AUROC
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic Surgery Cohort: Adults undergoing elective laparoscopic major abdominal surgery under general anesthesia at a single academic hospital. Each participant may receive up to two standardized 250-mL crystalloid fluid challenges (pre- and post-pneumoperitoneum). SVV and PVI are recorded around each bolus; no assignment or experimental treatment.
  Interventions: Device: Stroke Volume Variation (SVV) monitoring; Device: Pleth Variability Index (PVI) monitoring

INTERVENTIONS:
Device: Stroke Volume Variation (SVV) monitoring — Non-investigational physiologic monitoring. SVV derived from the invasive arterial pressure waveform using a commercially available platform. Used as an index test; values recorded immediately before and ~3 minutes after a standardized 250-mL crystalloid bolus at up to two time points (pre- and post-pneumoperitoneum). Readings are masked to clinicians; operation per usual care.
  Other Names: SVV; Arterial pressure waveform analysis; FloTrac; EV1000; HemoSphere; Edwards Lifesciences
Device: Pleth Variability Index (PVI) monitoring — Non-investigational pulse-oximetry-derived index. PVI obtained from a commercial monitor. Used as a paired index test; values recorded immediately before and ~3 minutes after each 250-mL crystalloid bolus (up to two time points). Readings masked; monitor used within standard care.
  Other Names: PVI; Pleth variability Index; Pulse oximetry-derived variability; Masimo; Radical-7

SUMMARY:
This study will compare two operating-room monitors-stroke volume variation (SVV, from the arterial line) and the Pleth Variability Index (PVI, from the pulse oximeter)-to see which one more accurately predicts whether giving a small fluid bolus will improve the heart's pumping during laparoscopic major abdominal surgery. Adults having elective surgery under general anesthesia will receive two small, timed 250-mL crystalloid infusions as part of routine care (one before and one after creation of the pneumoperitoneum). The research team will record SVV and PVI values just before and three minutes after each infusion while keeping these readings hidden from the clinicians so that usual care is not changed. No experimental drugs or devices are used. The main goal is to learn which index better identifies "fluid responsiveness," so future care can be safer and more consistent. Potential risks are minimal and relate to the small fluid boluses (temporary changes in blood pressure or heart rate); the test stops if the anesthesiologist has any safety concerns. There is no direct benefit to participants, but results may help guide fluid therapy for similar patients in the future. The study is being conducted at a single academic hospital in the Republic of Korea and plans to enroll about 300 adults.

DETAILED DESCRIPTION:
Background and rationale. Goal-directed fluid therapy during laparoscopic major abdominal surgery remains variable because dynamic preload indices perform inconsistently under pneumoperitoneum and positional changes. Stroke Volume Variation (SVV, derived from the arterial pressure waveform) and the Pleth Variability Index (PVI, derived from the pulse oximeter) are both widely available and non-drug, non-investigational monitors. A head-to-head, paired accuracy study using standardized fluid challenges can clarify which index better identifies fluid responsiveness in this setting.

Objectives. Primary: Compare the diagnostic accuracy (area under the ROC curve, AUROC) of SVV vs PVI for predicting fluid responsiveness to a small crystalloid bolus during laparoscopic major abdominal surgery.

Key secondary objectives: (1) determine optimal decision thresholds and report sensitivity, specificity, predictive values, and likelihood ratios; (2) compare calibration and classification performance (Youden index, net reclassification); (3) assess effect modification by pneumoperitoneum status, body mass index, ventilation parameters, and vasoactive use; (4) describe peri-bolus hemodynamic changes.

Design and setting. Prospective, single-center, paired diagnostic-accuracy cohort. Adults undergoing elective laparoscopic major abdominal surgery under general anesthesia are enrolled. Each participant undergoes up to two standardized 250-mL crystalloid fluid challenges delivered over ~3 minutes at two time points when feasible: (A) before insufflation and (B) after establishment of pneumoperitoneum at a hemodynamic steady state. Because both indices are recorded around the same fluid challenges, each participant serves as his/her own control.

Index tests. SVV (from the arterial pressure monitor) and PVI (from the pulse-oximetry monitor) are captured immediately before ("pre-bolus") and at ~3 minutes after each bolus. Index values are recorded by trained research staff and kept masked from anesthesia clinicians to avoid influencing usual care.

Reference standard and definition of fluid responsiveness. The reference standard is change in stroke volume index (SVI) or cardiac index derived from arterial pulse contour analysis. Fluid responsiveness is defined a priori as a ≥10% increase in SVI after the 250-mL bolus. Sensitivity analyses will use a 15% threshold and will repeat analyses with cardiac index. If signal quality is inadequate or a clinical safety concern arises, the test is aborted and data flagged.

Anesthesia and peri-bolus standardization. Ventilation is volume-controlled with tidal volume ~6-8 mL/kg predicted body weight and PEEP according to institutional practice; settings and pneumoperitoneum pressure/position are recorded. Vasoactive drugs and additional fluids are allowed as clinically indicated but are time-stamped; fluid challenges for research are not given when active titration of vasoactives makes a stable baseline impossible.

Participants. Inclusion: adults (≥18 years), ASA I-III, elective laparoscopic major abdominal surgery, arterial line in place, informed consent. Exclusion: clinically significant arrhythmia (e.g., atrial fibrillation with irregular R-R), severe valvular disease, intracardiac shunts, pregnancy, severe right-heart failure, inability to obtain reliable arterial or plethysmographic waveforms, or any condition in which a fluid challenge is judged unsafe by the anesthesiologist.

Outcomes. Primary outcome: AUROC of SVV vs PVI for predicting fluid responsiveness. Secondary outcomes: sensitivity/specificity at prespecified thresholds (e.g., SVV 12-13%, PVI 13-15%), decision-curve analysis, subgroup AUROC by pneumoperitoneum status, and immediate hemodynamic responses (MAP, HR).

Sample size and power. The study plans to enroll ~300 adults, yielding up to ~600 evaluable fluid challenges. Assuming a fluid-responsive rate of ~40%, this sample provides >80% power to detect a paired AUROC difference of ~0.08-0.10 between SVV and PVI at α=0.05 using DeLong's test with clustering by subject.

Statistical analysis. ROC curves for SVV and PVI are constructed using clustered bootstrap resampling at the patient level (≥2000 replicates). AUROCs are compared with paired DeLong tests. Threshold performance metrics include exact 95% CIs with patient-clustered bootstrap. Mixed-effects logistic regression (random intercept for patient) will estimate adjusted odds of fluid responsiveness per unit change of each index; prespecified covariates include pneumoperitoneum status, BMI, tidal volume per kg, PEEP, and vasoactive use. Missing index or reference values are minimized; if >5% are missing, multiple imputation will be performed in sensitivity analyses. All analyses follow a prespecified statistical analysis plan.

Safety and risk/benefit. Risks relate to small fluid boluses (transient blood pressure or heart-rate changes, fluid accumulation in vulnerable patients). The bolus is withheld or stopped for any safety concern. No experimental drugs or investigational devices are used; all monitors are standard of care. Participants are unlikely to benefit directly, but the results may improve future intraoperative fluid management.

Confidentiality and data handling. Data are captured on a secure electronic case-report form with coded identifiers. Only the research team has access. Results will be presented in aggregate without personal identifiers and disseminated in peer-reviewed venues.

Regulatory status. This is not an FDA-regulated drug or device investigation and is conducted under institutional review board approval at a single academic hospital in the Republic of Korea.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* ASA physical status I-III
* Elective laparoscopic major abdominal surgery under general anesthesia
* Arterial line in place for clinical care
* Able to provide informed consent
* Arterial and plethysmographic waveforms adequate for measurement

Exclusion Criteria:

* linically significant arrhythmia (e.g., atrial fibrillation with irregular R-R)
* Severe valvular heart disease or intracardiac shunt
* Pregnancy
* Severe right-heart failure or condition where a fluid bolus is unsafe
* Ongoing hemodynamic instability requiring rapid vasoactive titration at assessment
* Persistently unreliable arterial/pleth signals despite optimization
* Any situation the anesthesiologist judges that the fluid challenge is unsafe

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults undergoing elective laparoscopic major abdominal surgery at a single academic hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Area under the ROC curve (AUROC) of stroke volume variation (SVV) and Pleth Variability Index (PVI) for predicting fluid responsiveness to a 250-mL crystalloid bolus | Intraoperative: from the pre-bolus baseline to ~3 minutes after each standardized 250-mL crystalloid bolus (up to two episodes per participant: before and after pneumoperitoneum).
  Index tests: pre-bolus SVV (arterial waveform-derived) and PVI (pulse-oximetry-derived). Reference standard: fluid responsiveness defined as a >=10% increase in stroke volume index measured about 3 minutes after the 250-mL crystalloid bolus using arterial pulse contour analysis. ROC curves will be built for SVV and PVI to discriminate responders vs non-responders; AUROCs will be compared with a paired DeLong test with patient-level clustering. Unit: AUROC (0-1; higher indicates better discrimination).

SECONDARY OUTCOMES:
Sensitivity of prespecified SVV thresholds for predicting fluid responsiveness | Intraoperative: pre-bolus baseline to about 3 minutes after each 250 mL bolus (up to two boluses).
  Proportion of fluid challenges in which SVV > 13% correctly identifies fluid responsiveness (≥10% increase in stroke volume index after a 250 mL bolus).Unit of Measure: Percent of fluid challenges (%)
Specificity of prespecified SVV thresholds for predicting fluid responsiveness | Intraoperative: pre bolus baseline to about 3 minutes after each 250 mL bolus (up to two episodes per participant).
  Proportion of fluid challenges in which SVV ≤ 13% correctly identifies non-responsiveness.
  Unit of Measure: Percent of fluid challenges (%)
Sensitivity of prespecified PVI threshold for predicting fluid responsiveness | Intraoperative: pre bolus baseline to about 3 minutes after each 250 mL bolus (up to two episodes per participant).
  Description: Proportion of fluid challenges in which PVI > 15% correctly identifies fluid responsiveness (≥10% increase in stroke volume index).
  Unit of Measure: Percent of fluid challenges (%)
Specificity of prespecified PVI threshold for predicting fluid responsiveness | Intraoperative: pre bolus baseline to about 3 minutes after each 250 mL bolus (up to two episodes per participant).
  Proportion of fluid challenges in which PVI ≤ 15% correctly identifies non-responsiveness.
  Unit of Measure: Percent of fluid challenges (%)
Optimal cutoffs for SVV using Youden index | Intraoperative: pre bolus to about 3 minutes post bolus.
  Data-driven SVV threshold (%) that maximizes the Youden index (sensitivity + specificity - 1) for predicting fluid responsiveness.
  Unit of Measure: Percent (%)
Optimal cutoffs for PVI using Youden index | Intraoperative: pre bolus to about 3 minutes post bolus.
  Data-driven PVI threshold (%) that maximizes the Youden index for predicting fluid responsiveness.
  Unit of Measure: Percent (%)
Percent change in stroke volume index after a fluid bolus | Intraoperative: pre bolus baseline to about 3 minutes after each 250 mL bolus.
  Percent change in stroke volume index from pre-bolus baseline to about 3 minutes after each 250 mL bolus; subgroup analyses will compare periods before vs. after pneumoperitoneum. Unit of Measure: Percent change (%)
Change in mean arterial pressure after fluid challenge | Intraoperative: pre bolus to about 3 minutes post bolus.
  Absolute change in mean arterial pressure (mmHg) from pre-bolus baseline to about 3 minutes after each 250 mL bolus.
  Unit of Measure: Millimeters of mercury (mmHg)
Change in heart rate after fluid challenge | Intraoperative: pre bolus to about 3 minutes post bolus.
  AAbsolute change in heart rate (beats per minute) from pre-bolus baseline to about 3 minutes after each 250 mL bolus.
Incidence of any predefined hemodynamic adverse event within 10 minutes of a study bolus | From bolus start to 10 minutes after each bolus during surgery.
  Number of participants experiencing at least one predefined hemodynamic adverse event (hypotension requiring vasopressor, tachycardia requiring treatment, new arrhythmia, etc.) within 10 minutes after each study bolus, divided by the total number of participants. Unit of Measure: Percent of participants (%)

CONTACTS AND LOCATIONS:
Overall Officials: Cheolhyeong Lee, MD, PhD, Principal Investigator — Wonkwang University School of Medicine Hospital
Locations (1):
- Wonkwang University School of Medicine Hospital, Iksan, Jeollabuk-do, South Korea